CLINICAL TRIAL: NCT03693768
Title: Motivational Encouragement With Networks (MEN) for Healthy Eating Activity Resting Together (HEART) Health Study
Acronym: MEN 4 HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Larrell L Wilkinson, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300001419
Record Dates: First submitted 2018-06-21; First posted 2018-10-03 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-06

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health coaching ARM (Experimental): Participants in this ARM will undergo health coaching for 4 months.
  Interventions: Behavioral: Health coaching

INTERVENTIONS:
Behavioral: Health coaching — Health coaching

SUMMARY:
The purpose of this research study is to determine if a health coaching intervention that includes exercise, good dietary habits, and good relaxation methods helps overweight men improve health and lose weight. The investigator's hope is to enroll 30 men in this research study.

DETAILED DESCRIPTION:
Health coaching helps patients gain the knowledge, skills, tools and confidence to become active participants in their care so that they can reach self-identified health goals. Health coaching: 1) provides self-management support, 2) bridges gaps between health professionals and patients, 3) helps patients navigate the health care system, 4) offers emotional support, and 5) serves as a continuity figure. The intervention will consist of tailored health coaching, goal setting, and behavioral contracting for healthy actions to create a supportive context for participants that supports health promoting behaviors (HPBs), with efforts to enhance HPB reinforcement through established networks. After baseline assessment, the men will participate in a 45-minute educational meeting with the principal investigator (PI) to discuss self-reported measures from baseline instruments and the importance of health promoting behaviors (HPBs) to overall heart health. Afterwards, a research study team (research trained undergraduate and graduate student assistants) will perform case management and health advisement (bi-weekly continuity phone calls 2x / month) to support protocol adherence and tracking of participant goals over a period of 120 days. The research team will be guided by a coaching manual created for the purposes of the study. The M for H study will also create and provide health-oriented emails (2x / week), daily tracking text messaging on weekdays, monthly face-to-face coaching group meetings during community-based organization (CBO) set times (i.e. meetings, events), and access to an optional social media platform supporting peer interactions. After 120 days, participants will be reassessed to determine impacts related physical activity (PA) measures, knowledge, attitudes, & practices (KAPs), and interviewed to discuss M for H feasibility and acceptability. The targeted outcome for the 120 day period will be improvement toward the performance of >150 minutes of moderate to vigorous physical activity accumulated as indicated by accelerometry, increase in distance walked during a six (6) minute walk test, and improvement in theoretical construct measures indicative of performance of HPBs among participants.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible if they are African American (AA) men:

* 45 - 75 years of age at initial enrollment in the study
* Overweight (BMI 25 - 29.99)
* Obese (BMI 30 - 44.99)
* Sufficiently inactive (i.e. self-report accumulating <90 minutes/week of moderate or vigorous physical activity)
* Categorized as low or moderate risk in accordance with American College of Sports Medicine (ACSM) guidelines for pre-exercise screening

Exclusion Criteria:

* Younger than 45 years
* Not able to speak or read English
* Life expectancy of less than 1 year
* Categorization of high risk in accordance with ACSM guidelines
* Identified by one's primary care clinician as unable to follow instructions because of physical or cognitive disability
* Psychiatric illness
* Other unidentified reasons as determined by the investigators

Ages: 45 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | 4 months
  Change in weekly physical activity minutes accumulated from baseline measures assessed by employing accelerometry.

SECONDARY OUTCOMES:
Change in fruit / vegetable intake | 4 months
  Change in daily fruit and vegetable intake from baseline measures assessed by questionnaire (food log journal).
Change in sleep hours nightly | 4 months
  Change in nightly sleep hours measured nightly from baseline measures assessed by questionnaire.

OTHER OUTCOMES:
Change in Weight Measurement | 4 months
  Change in weight (lbs.) from baseline measure assessed via Omron scale.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No